CLINICAL TRIAL: NCT02747524
Title: Haiti Rural School Feeding Study: Effects of Vita Mamba on Anemia and Hemoglobin Concentrations
Brief Title: Haiti Rural School Feeding Study: Effect of Vita Mamba on Anemia and Hemoglobin Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201207037
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vita Mamba (Experimental): Nutrient fortified peanut butter paste for 26 weeks.
  Interventions: Other: Vita Mamba peanut butter paste
- Control (No Intervention)

INTERVENTIONS:
Other: Vita Mamba peanut butter paste
  Arms: Vita Mamba

SUMMARY:
This study applied a matched cluster, controlled design, using community cluster as the unit of randomization. Communities were first matched during the formative research phase and randomized into treatment (Vita Mamba + deworming) or control (deworming) groups, using a simple experimental 1:1 design. The principal investigator generated the random allocation sequence and assigned the cluster to groups. Children were followed longitudinally for Hb concentration and anthropometric measures were taken at baseline (November 2014) and endline (June 2015). Parents were surveyed at baseline for household-level socioeconomic and demographic information; environmental conditions including water, hygiene, and sanitation; and child diet and morbidities.

All children in the intervention schools received the Vita Mamba once per school day from November 2014 to June 2015, for approximately 26 weeks. Children in both groups received Albendazole at baseline in November 2014. Compliance was monitored by teachers and tracked by collection of empty packages. Lessons learned from another school feeding trial by the study team were applied to increase compliance such as opening the packages for the children immediately prior to consumption to discourage selling or sharing later with family members. Vita Mamba was developed for the urban school trial by the research team with representatives from Edesia (a US-based nonprofit manufacturer of ready-to-use foods with expertise in research and development) and Nutriset (the parent company in the PlumpyField network). Meds & Food for Kids, a nonprofit manufacturer of ready-to-use foods in Haiti using locally produced peanuts, produced the Vita Mamba for this trial. Vita Mamba (50 g) contains 260 kcal and meets >75% of the Recommended Dietary Allowance (RDA) for critical micronutrients (S1 Table).

ELIGIBILITY:
Inclusion Criteria:

* registration in the study school for 2014-2015 calendar; good health (no fever, congenital health condition, or peanut or soy allergy); and not severely malnourished (weight-for-height [WHZ] <-3)

Exclusion Criteria:

* fever, congenital health condition, or peanut or soy allergy; severely malnourished (weight-for-height [WHZ] <-3)

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
hemoglobin concentration | 26 weeks

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Palacios AM, Freeland-Graves JH, Dulience SJ, Delnatus JR, Iannotti LL. Differences in factors associated with anemia in Haitian children from urban and rural areas. PLoS One. 2021 Apr 6;16(4):e0247975. doi: 10.1371/journal.pone.0247975. eCollection 2021. PMID 33822795